CLINICAL TRIAL: NCT05801146
Title: A Double-blind, Randomized, Parallel, Active-controlled, Non-inferiority, Phase III Clinical Trial to Compare the Efficacy and Safety of HG102 Versus Botox® in Subjects With Moderate to Severe Glabellar Lines
Brief Title: Evaluate the Safety and Efficacy of HG102 as Compared to Botox® in Subject With Moderate to Severe Glabellar Lines
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HG-102GL-PIII-01
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin type A(HG102) (Experimental)
  Interventions: Drug: Botulinum Toxin Type A Injection [HG102]
- Botulinum toxin type A(Botox®) (Active Comparator)
  Interventions: Drug: Botulinum Toxin Type A Injection [Botox]

INTERVENTIONS:
Drug: Botulinum Toxin Type A Injection [HG102] — Single administration, Day 0, 20 units
  Other Names: HG102
  Arms: Botulinum toxin type A(HG102)
Drug: Botulinum Toxin Type A Injection [Botox] — Single administration, Day 0, 20 units
  Other Names: Botox®
  Arms: Botulinum toxin type A(Botox®)

SUMMARY:
To evaluate the efficacy and safety of HG102 for moderate to severe Glabellar Lines, non-inferiority compared to Botox® was confirmed and safety was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that fit all of the criteria below were selected for this clinical trial.

  1. Male and female adults from 19 to 65 years old at the time of screening
  2. Person with moderate or severe glabellar lines and have received Grade 2-3 according to Physician's Rating Line Severity at maximum frown
  3. Person who understands and can comply to the process and visiting schedule of this clinical study
  4. Person who gave spontaneous written consent to participate in this clinical study

Exclusion Criteria:

* Subjects that fit any of the criteria below were excluded from this clinical trial.

  1. Person with infection, skin disease, or scar on forehead
  2. Person with symptoms of facial palsy or blepharoptosis
  3. Person with allergies or hypersensitive reaction history to the ingredients in the investigational product (botulinum toxin formula, serum albumin, etc.)
  4. Person who were administered with similar medication within 12 weeks (botulinum toxin type A medication) or 16 weeks (botulinum toxin type B medication)
  5. Pregnant and breast-feeding women, men and women in the childbearing age who are planning to get pregnant during the clinical study period, or do not agree to the suitable contraceptive methods
  6. Person who participated in another clinical trial, or were given medication for other clinical trials within 4 weeks from screening of 5 times the half-life, which period may be longer
  7. Other person who the investigator judges as inappropriate for the clinical trial

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Responder rate of improvement in glabellar lines with Physician's rating line severity | Baseline to week 4
  Improvement rate of glabellar lines at maximum frown with Physician's rating line severity at 4 weeks post injection

SECONDARY OUTCOMES:
Responder rate of improvement in glabellar lines with Physician's rating line severity | Baseline to week 8, 12, 16
  Improvement rate of glabellar lines at maximum frown with investigator's photo assessment at 8, 12, 16 weeks post injection
Responder rate of improvement in glabellar lines with investigator's photo assessment | Baseline to week 4, 8, 12, 16
  Improvement rate of glabellar lines at rest with Physician's rating line severity at 4, 8, 12, 16 weeks post injection
Responder rate of improvement in glabellar lines with investigator's photo assessment | Baseline to week 4, 8, 12, 16
  Improvement rate of glabellar lines at rest with investigator's photo assessment at 4, 8, 12, 16 weeks post injection
Independent photo evaluator-rated improvement rate of glabellar lines at rest | Baseline to week 4, 8, 12, 16
Responder rate of improvement in glabellar lines with Subject's improvement assessment | Baseline to week 4, 8, 12, 16
  Improvement rate of glabellar lines with Subject's improvement assessment at 4, 8, 12, 16 weeks post injection
Participant-rated satisfaction after treatment | Baseline to week 4, 8, 12, 16
  Subject's satisfaction rate of improvement in glabellar lines at 4, 8, 12, 16 weeks post injection

CONTACTS AND LOCATIONS:
Locations (1):
- Hugel, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No